CLINICAL TRIAL: NCT01792713
Title: Randomisierte, Doppelblinde, Plazebo-kontrollierte Prüfung Zum Nachweis Der Wirksamkeit Und Der Lokalen Verträglichkeit Einer 2%Igen Sertaconazol-Crème Bei Patienten Mit Atopischer Dermatitis (Abridged)
Brief Title: Sertaconazole 2% Cream to Improve Symptoms Associated With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spirig Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E550-PRU-2012; 2012-003954-95 (EudraCT Number)
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Skin Alterations Associated With Atopic Dermatitis
Keywords: Skin alterations; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — sertaconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sertaconazole 2% cream (Active Comparator): 2x daily treatment with Sertaconazole 2% cream for 4 weeks, 2 weeks follow-up
  Interventions: Drug: Sertaconazole 2% cream
- Placebo Arm (Placebo Comparator): 2x daily treatment with Placebo cream for 4 weeks, 2 weeks follow-up
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sertaconazole 2% cream
  Arms: Sertaconazole 2% cream
Drug: Placebo
  Arms: Placebo Arm

SUMMARY:
Investigation aimed to explore the efficacy of a topical Sertaconazole cream 2% in patients with skin alterations associated with atopic dermatitis

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Atopic Dermatitis Patients with SCORing Atopic Dermatitis (SCORAD) ≤ 40
* Atopic lesion localisation: arms; additional legs, neck

Exclusion Criteria:

* SCORAD > 40
* Unstable, uncontrolled medical status (e.g. active systemic or topical infection)
* Active immunosuppression or cancer
* Narcotics- or Alcohol abuse
* Participation in another clinical trial until one month prior inclusion
* Known allergies against an ingredient of the investigational medicinal product
* Different periods of grace for certain pre-treatments, e.g. topical corticosteroids, immune modulating drugs
* Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-02; Primary Completion 2013-09 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in Patient Global Assessment (PGA) | day 1, day 28

SECONDARY OUTCOMES:
Change in Eczema Area and Severity Index (EASI) | day 1, day 28
Change in Dermatology Life Quality Index (DLQI) | d1, d28
Change in Patient Benefit Index (PBI) | day 1, day 28

OTHER OUTCOMES:
Change in Transepidermal water loss (TEWL) | d1, d14, d28, d42

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Universitätsmedizin Charité Berlin, Abteilung für Dermatologie und Allergologie, Berlin
  - Universitätsklinikum Münster, Klinik für Hautkrankheiten, Münster

REFERENCES:
- [Derived] Stander S, Metz M, Ramos F MH, Maurer M, Schoepke N, Tsianakas A, Zeidler C, Luger TA. Anti-pruritic Effect of Sertaconazole 2% Cream in Atopic Dermatitis Subjects: A Prospective, Randomized, Double-blind, Vehicle-controlled, Multi-centre Clinical Trial of Efficacy, Safety and Local Tolerability. Acta Derm Venereol. 2016 Aug 23;96(6):792-6. doi: 10.2340/00015555-2268. PMID 26527564